CLINICAL TRIAL: NCT01256853
Title: A Phase I, Dose Escalation Trial of Recombinant Modified Vaccinia Ankara (MVA)-Based Vaccine Encoding Epstein-Barr Virus Target Antigens
Brief Title: Modified Vaccinia Ankara (MVA) Vaccine Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CCTU, Comprehensive Clinical Trial Unit, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAC002
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Last update posted 2011-12-22 (Estimated); Status verified 2011-12

CONDITIONS: Nasopharyngeal Neoplasms; Epstein-Barr Virus Infections
Keywords: histologically confirmed EBV+ NPC patients
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Epstein-Barr Virus Infections | interventions — MVA vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MVA Vaccine (Experimental)
  Interventions: Drug: MVA Vaccine

INTERVENTIONS:
Drug: MVA Vaccine — The starting dose will be 5 x 107 plaque forming units (pfu) given by intradermal vaccination. Cohorts of three patients will receive escalating doses of the vaccine (100%, 100%, 67% and 50%). The dose escalation scheme is 5 x 107 pfu, 1 x 108 pfu, 2 x 108 pfu, 3.3 x 108 pfu, 5 x 108pfu. This will be dependant on toxicity.

SUMMARY:
This is a phase I, dose escalation trial of MVA-EBNA1/LMP2 vaccine across a pre-defined range of doses in patients in remission having had an EBV+ nasopharyngeal carcinoma (NPC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed NPC, in which the presence of EBV within the malignant cells has been demonstrated by (1) EBER (EBV early RNA) in situ hybridisation in more than 50% of the malignant cells, or (2) undifferentiated or poorly differentiated carcinoma histology in association with a raised serum titer of IgA to EBV VCA.
* Patients in remission from disease, ie complete response (CR) or unconfirmed complete response (CRu).
* Completion of standard therapy for malignancy at least 12 weeks before trial entry.
* Written informed consent and the ability of the patient to co-operate with treatment and follow up must be ensured and documented.
* Age greater than 18 years.
* World Health Organisation (WHO) performance status of 0 or 1
* Life expectancy of at least 4 months.
* Haematological and biochemical indices (these measurements must be performed within 28 days prior to the patient going on study):

  * Haemoglobin (Hb) > 10.0 g/dl
  * Lymphocytes > 1.0 x 109/L (or above the lower limit of normal range of institutional laboratory)
  * Neutrophils ≥ 1.5 x 109/L
  * Platelets (Plts) ≥ 100 x 109/L
  * baseline liver function tests :
  * Serum bilirubin ≤ 1.5 x upper normal limit
  * Serum alkaline phosphatase, alanine amino-transferase (ALT) and/or aspartate amino-transferase (AST) < 1.5 x ULN.
  * baseline renal function test:
  * calculated creatinine clearance > 50ml/min Female patients of child-bearing potential are eligible, provided they have a negative pregnancy test prior to enrolment and agree to use appropriate medically approved contraception during the study up to six months after the last vaccination.
* Male patients must agree to use appropriate medically approved contraception during the study up to six months after the last vaccination.

Exclusion Criteria:

* Receiving current chemotherapy or radiotherapy, or received within 12 weeks of trial entry.
* Known chronic active infection with Hepatitis B, Hepatitis C or Human Immunodeficiency Virus (HIV).
* Current active autoimmune disease.
* Current active skin diseases requiring therapy (psoriasis, eczema etc).
* Ongoing active infection.
* History of anaphylaxis or severe allergy to vaccination.
* Allergy to eggs or egg products.
* Previous myeloablative therapy followed by an autologous or allogeneic haematopoietic stem cell transplant.
* Patients who have had a splenectomy or splenic irradiation, or with known splenic dysfunction.
* Receiving current immunosuppressive medication, including corticosteroids.
* Pregnant and lactating women.
* Ongoing toxic manifestations of previous treatment. Exceptions to this are alopecia or certain Grade 1 toxicities which in the opinion of the Investigator and Cancer Research UK should not exclude the patient.
* Major thoracic and/or abdominal surgery in the preceding four weeks from which the patient has not yet recovered.
* Patients with any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.
* Concurrent congestive heart failure or prior history of class III/ IV cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To determine safety and to characterise the toxicity profile of MVA-EBNA1/LMP2 vaccine | 4 years

SECONDARY OUTCOMES:
To describe changes in the frequency of functional T-cell responses to MHC class I and II-restricted epitopes within EBNA1 and LMP2 in peripheral blood at sequential time-points before, during and up to nine months after the vaccination course. | 4 years
To assess changes in levels of EBV genome levels in plasma | 4 Years

CONTACTS AND LOCATIONS:
Overall Officials: Anthony TC Chan, MD, FRCP, Principal Investigator — Department of Clinical Oncology, The Chinese University of Hong Kong
Locations (1):
- Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong, Hong Kong